CLINICAL TRIAL: NCT03758898
Title: The Effect of Chest Physiotherapy After Bariatric Surgery on Pulmonary Functions, Functional Capacity and Quality of Life
Brief Title: The Effect of Chest Physiotherapy After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Asst. Prof. Ph.D., Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBU11.2018
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Bariatric Surgery Candidate; Pulmonary Disease
Keywords: Bariatric surgery; Chest physiotherapy; Pulmonary functions; Quality of life
MeSH Terms: conditions — Lung Diseases | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The patients were randomised using randomisation software and divided into two groups each comprising 74 patients. Chest physiotherapy and mobilisation was applied to the patients in the first group, and only mobilisation was applied to the patients in the second group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Chest physiotherapy and mobilisation were applied on the patients for 4 days. The treatment of the patients was started on the first postoperative day and continued until the postoperative 4th day.
  Interventions: Other: Treatment; Other: Group 2
- Group 2 (Placebo Comparator): only mobilisation was applied to the patients in the second group
  Interventions: Other: Treatment; Other: Group 2

INTERVENTIONS:
Other: Treatment — Chest physiotherapy and mobilization were applied twice a day, 8 times in total.
Other: Group 2 — Only mobilization was applied twice a day, 8 times in total.

SUMMARY:
The aim of this study was to investigate the effect of chest physiotherapy applied to patients undergoing bariatric surgery on pulmonary functions, dyspnea levels, functional capacity and quality of life.

DETAILED DESCRIPTION:
This randomized, controlled trial, was designed, conducted, and reported in accordance with the standards of The CONSORT (Consolidated Standards of Reporting Trials) Statement. The patients were randomised and divided into two groups each comprising 74 patients. Chest physiotherapy and mobilisation was applied to the patients in the first group, and only mobilisation was applied to the patients in the second group. The treatment of the patients was started on the first postoperative day and continued until the postoperative 4th day. Chest physiotherapy and mobilization were applied twice a day, 8 times in total. The following parameters were evaluated preoperative and postoperative:arterial blood gas, oxygen saturation, respiratory function test for pulmonary functions, pulmonary artery pressure for pulmonary hypertansion, Borg dyspnea score for severity of dyspnoea, 6-minute walk test for functional capacity, Nottingham health profile for quality of life.

Chest physiotherapy consisted of postural drainage (30-45 degree eleve), breathing exercises (deep breathing, diaphragm breathing, active breathing techniques cycle) and coughing techniques (huffing, controlled coughing, manual assisted coughing). In the chest physiotherapy program, diaphragmatic respiration, constrictive lip respiration, segmental respiration, incentive spirometry and coughing were performed on the 1st postoperative day. All respiratory exercises were repeated twice a day and percussion was added on the 2nd postoperative day. All respiratory exercises and percussion were repeated 2 times a day until the discharge of the post op day 4 until discharge, and the work with incentive spirometry was removed per hour. Patients were mobilized as early as possible by the physiotherapist. The patients in both groups were instructed to sit out of bed and stand up on the first postoperative day, walk 45 m in the corridor on the second day, walk freely (approximately 150-300 m) on the third and the fourth days.

All operations were laparoscopic, sleeve gastrectomy or Roux-en Y gastric bypass (21). Routine anesthesia was performed with desflurane and remifentanil. In all procedures, patients were treated with the split upward position (French position) and a semi-reclining position (anti-Trendelenburg position). All patients received prophylaxis against deep vein thrombosis for 2 weeks with pneumatic compression stocking and subcutaneous low molecular weight heparin. Perioperative antibiotics (cefazolin 2 g) were also routinely administered. The patients were discharged on the fourth postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* obese and morbidly obese patients
* aged between 30 and 50 years

Exclusion Criteria:

* previous obesity surgery
* presence of chronic respiratory disease
* renal / hepatic dysfunction
* malignant hyperthermia
* regular alcohol
* smoking and drug use
* pregnancy.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Body mass index | 1 minute
  BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The National Institutes of Health (NIH) now defines normal weight, overweight, and obesity according to BMI rather than the traditional height/weight charts. Overweight is a BMI of 27.3 or more for women and 27.8 or more for men. Obesity is a BMI of 30 or more for either sex (about 30 pounds overweight). A very muscular person might have a high BMI without health risks.

SECONDARY OUTCOMES:
Functional capacity: 6 minute walk test | 5 minutes
  The subjects were instructed to walk as far as possible in six minutes in an enclosed 50-m long hospital corridor. Standardized encouragement was given in every 30 s. The maximum distance covered at the end of the test was recorded
Dispnea: Borg scale | 6 minutes
  Breathlessness and fatigue perception were determined using a 10-point modified Borg scale during the six minute walking test. Total score is 10 points. "This is a scale that asks you to rate the difficulty of your breathing. It starts at number 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal. How much difficulty is your breathing causing you right now?" 0 better, 10 worst point mean.
Quality of Life profile: Nottingham Health Profile | 8 minutes
  Nottingham Health Profile (NHP) was used to determine quality of life of the participants. NHP is a general health status scale (health-related quality of life), which aims to measure a patient's perceived emotional, social and physical health status. This scale consists of 38 items formed as yes-no questions that cover 6 subscales of the quality of life. These six subscales are sleep (5 item), energy level (3 item), emotional status (9 item), social isolation (5 item), physical mobility (8 item) and pain (8 item). Each section is scored from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Tomri̇s Duymaz, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Tomri̇s Duymaz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No